CLINICAL TRIAL: NCT00211562
Title: Reduction of Body Weight in Olanzapine Treated Schizophrenia Patients by Adjunctive Supplementation of Antioxidants (Vitamins E + C) Plus Omega-3 Fatty Acids
Brief Title: Adjunctive Supplementation of Antioxidants (Vitamins E + C) Plus Omega-3 Fatty Acids
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Augusta University (Other)
Collaborators: Eli Lilly and Company (Industry); Medical Service Line ABRC (Unknown); US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Omega-3 Fatty Acids
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2012-10-24 (Estimated); Status verified 2012-10

CONDITIONS: Schizophrenia
Keywords: weight gain; weight gain supplementation; antioxidants; olanzapine
MeSH Terms: conditions — Schizophrenia; Weight Gain | interventions — Olanzapine; Docosahexaenoic Acids

ARMS (3):
- Olanzapine (Active Comparator)
  Interventions: Drug: Olanzapine, Omega 3, Vitamin E+C
- Omega 3 (Active Comparator)
  Interventions: Drug: Olanzapine, Omega 3, Vitamin E+C
- Vitamin E +C (Active Comparator)
  Interventions: Drug: Olanzapine, Omega 3, Vitamin E+C

INTERVENTIONS:
Drug: Olanzapine, Omega 3, Vitamin E+C — No adverse event nor SAE noted.

SUMMARY:
This research study helps to demonstrate that adding vitamins and fats (nutritional supplements) to a diet will help reduce body weight and improve the lipid profile. This will be done by examining the body weight and chemicals in the blood. The chemicals are the result of the brain using the fat that subjects eat in their diet. Some medications may also change the amount of these chemicals in a person's blood.

DETAILED DESCRIPTION:
To demonstrate that supplementation of antioxidants and omega-3 fatty acids will improve clinical outcome including cognitive performance in olanzapine treated patients.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 55
* VA outpatient
* Diagnosis of schizophrenia by DSM-IV criteria
* Active treatment with olanzapine
* Medically healthy

Exclusion Criteria:

* Diagnosis of MR
* MMSE score of < 26
* Not on a stable dose of olanzapine

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2005-10; Primary Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
PANSS | 2003-2006
  Study completed in 2006. PI no longer with the institution. Study was closed accordingly to the HAC.
BMI | 2003-2006
  BMI match height and weight.
Blood samples | 2003-2006
  Samples analyzed, PI analyzed and published. PI no longer with the institution.

SECONDARY OUTCOMES:
Cognitive assessments | 2003-2006
  BACS assessment. Data analyzed and published by the PI.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Buckley, M.D., Principal Investigator — VA MC/Medical College of Georgia
Locations (1):
- VA Medical Center, Augusta, Georgia, United States

REFERENCES:
- [Background] Jones B, Basson BR, Walker DJ, Crawford AM, Kinon BJ. Weight change and atypical antipsychotic treatment in patients with schizophrenia. J Clin Psychiatry. 2001;62 Suppl 2:41-4. PMID 11232752
- See also: Related Info — http://www.ncbi.nlm.nih.gov